CLINICAL TRIAL: NCT05358925
Title: Online Psychoeducational Videos and Digital Assessments as a Method for Broadening Access to Care for Borderline Personality Disorder
Brief Title: Psychoeducational Videos and Digital Assessments for BPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Lois W. Choi-Kain, MD, Director, Gunderson Personality Disorder; Associate Professor of Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000892; 30053 (Other Grant/Funding Number: Brain and Behavior Research Foundation)
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; ecological momentary assessment; psychoeducation; neuropsychological feedback; symptom tracking
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: This study includes two randomization branching points: (1) BPD-related videos vs. non-BPD-related videos, and (2) receive neuropsychological feedback vs. not. At branching point (1), 2/3 of participants will be directed to the BPD-video condition, and 1/3 to the non-BPD-video condition. Only the participants in the BPD-video condition will be randomized to receive feedback or not (1/2 each condition). No non-BPD-video participants will receive feedback.
Masking Description: While the investigators will not explicitly inform participants of their condition, it will be apparent based on the content of the videos they receive and whether or not they receive feedback.
  The investigators and study staff will be aware of condition assignments in order to facilitate the delivery of the appropriate videos and the neuropsychological feedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BPD Videos and Feedback (Experimental): Ten daily 4-10 minute psychoeducational videos about BPD and personalized feedback about performance on neuropsychological tasks.
  Interventions: Other: Psychoeducational Videos; Other: Neuropsychological Feedback
- BPD Videos and No Feedback (Experimental): Ten daily 4-10 minute psychoeducational videos about BPD.
  Interventions: Other: Psychoeducational Videos
- Non-BPD Videos and No Feedback (Sham Comparator): Ten daily 4-10 minute educational videos about health-related topics other than BPD.
  Interventions: Other: Non-BPD-related Educational Videos

INTERVENTIONS:
Other: Psychoeducational Videos — A total of ten videos will be delivered daily Monday-Friday over approximately 2 weeks (days 1-15). The videos will each feature a mental health professional who is an expert in BPD explaining the topic in relatable language that can be understood by the general public. Each video will be approximately 4-10 minutes long, for a total of ~72 minutes of video. Videos will be shared via a hyperlink in a text message.
  The psychoeducational videos will cover the following topics: symptoms, basic factors about BPD, the naturalistic long term course of BPD, prevalence of BPD and its common comorbid disorders, key principles for recovery, available psychotherapeutic treatment options for BPD, common factors amongst treatments, medications, the interpersonal hypersensitivity model of BPD, and a review of the top 10 tips.
  Arms: BPD Videos and Feedback; BPD Videos and No Feedback
Other: Neuropsychological Feedback — In the second phase of the study, participants randomized to the Feedback condition will receive an email with a personalized summary of their symptom endorsement and neuropsychological performance. The feedback will include the relevant scores or sub-scores for each cognitive test (CPT, RMET, BEST, DST) from the first two time points. For each score and sub-score, there will be a description of the cognitive domain that the metric assesses (e.g., attention span in the CPT). The investigators will tailor the feedback to each participant's scores. The investigators may adjust the format or wording of the feedback based on participant responses (i.e., if a participant alerts the investigators that some wording is unclear or confusing). The investigators may also alter the feedback if they learn new information about the relevance or interpretability of these cognitive tests, as this is a growing field of research.
  Arms: BPD Videos and Feedback
Other: Non-BPD-related Educational Videos — The non-BPD-related educational videos will be matched in length and frequency to the BPD-related videos. These videos will discuss aspects of mental and physical health that are not related to BPD. Examples may include: nutrition and healthy eating, coping, self-compassion and self-care, stress and anxiety, depression, and healthy sleep habits.
  Arms: Non-BPD Videos and No Feedback

SUMMARY:
In this study, 100 adults who were recently diagnosed with borderline personality disorder (BPD) will be randomized to either receive educational videos about BPD or educational videos about other topics. All participants in both conditions will complete daily surveys about their emotions and social interactions, and they will respond to surveys and complete cognitive tests at 4 different time points. Some participants will receive feedback about their cognitive test performance, and others will not. The investigators are interested in learning about how accurate education about BPD and enhanced knowledge about cognitive abilities might help people manage their BPD symptoms. The investigators expect that participants who received psychoeducation about BPD will have lower levels of BPD and depressive symptoms than other participants, and that participants who received feedback on their cognitive tests will also have lower symptoms.

DETAILED DESCRIPTION:
In this study, 100 adults who were diagnosed with BPD within the past three months will be randomly assigned to receive psychoeducational videos (4-10 minutes each) about the development, symptoms, naturalistic trajectory, and treatment of BPD (2/3 of participants) or matched-length videos about non-BPD, health-related topics (1/3 of participants). One video will be delivered every business day for two weeks. Participants will respond to 5-minute surveys on their recent social interactions, their feelings of threat, connectedness, and aloneness, and will complete a 1-minute version of the Continuous Performance Test (CPT) and Digit Symbol Matching Test, every day for 30 days. Participants will complete additional full-length surveys and cognitive tests at 4 time points: baseline (Day 1), Time 2 (day 15), Time 3 (Day 30), and Follow-up (day 60). The primary outcome is BPD symptom severity, and the secondary outcome is depressive symptom severity. The investigators expect that BPD-focused psychoeducation and personalized neuropsychological feedback will each lead to separate, measurable reductions in BPD and depressive symptom severity. The investigators also expect that the relationship between psychoeducation and symptom reduction will be mediated by increased knowledge about BPD, and that the relationship between neuropsychological feedback and symptom reduction will be mediated by increased cognitive control.

ELIGIBILITY:
Inclusion Criteria:

* reliable access to a smartphone with a data plan for the duration of the study
* ability to speak and understand English
* age 18 years or older
* diagnosis of BPD within the past 6 months
* awake and able to complete EMA surveys between 9:00am and 9:00pm on most days
* located within the United States

Exclusion Criteria:

* cognitive disability that impedes ability to participate in the study
* current psychiatric symptoms that interfere with the individual's ability to provide consent or complete the research procedures (e.g., acute mania, acute psychosis, eating disorder threatening medical stability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Borderline Symptom List 23 (BSL-23) | Baseline (day 1), Time 2 (day 15), Time 3 (day 30), Follow-Up (day 60)
  Change (increase or decrease) in BSL-23 mean score (average score across all 23 items) at time 2, time 3, and follow-up, as compared to baseline. Minimum score = 0, maximum score = 4. A higher score indicates more severe BPD symptoms.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline (day 1), Time 2 (day 15), Time 3 (day 30), Follow-Up (day 60)
  Change (increase or decrease) in PHQ-9 total score at time 2, time 3, and follow-up, as compared to baseline. Minimum score = 0, maximum score = 27. A higher score indicates more severe depressive symptoms.

OTHER OUTCOMES:
Treatment History Questionnaire | Baseline (day 1), Follow-Up (day 60)
  Change between baseline and follow-up on the following metrics: A) Amount of treatment received in each of the following categories: individual therapy (# appointments per week for X weeks), group therapy (# months in group), day treatment (# days in program). B) Number of past psychiatric hospitalizations. C) History of BPD-specialized psychotherapy (yes/no).
  The minimum value is 0 for all questions on this questionnaire (e.g., 0 past hospitalizations). There is no maximum value for any question. A higher level of past engagement with mental health services may indicate a history of more severe psychopathology, or may indicate a greater level of access to mental health services, or a combination of these factors.
BPD Knowledge Assessment | Baseline (day 1), Time 2 (day 15), Follow-Up (day 60)
  Change (increase or decrease) in BPD Knowledge Assessment total score at time 2 and follow-up, as compared to baseline. This instrument is currently in development. A higher score will indicate a greater level of knowledge related to BPD.
Hospitalization Check-In | Time 2 (day 15) and Time 3 (day 30)
  Number of patients who have been hospitalized.
McLean Assessment of Rejection Sensitivity (MARS) | Baseline (day 1), Follow-Up (day 60)
  Change (increase or decrease) in MARS total score between baseline and follow-up. Minimum score = 11, maximum score = 55. A higher score indicates a greater sensitivity to rejection.
3-Item Loneliness Scale (LS-3) | Baseline (day 1), Time 2 (day 15), Time 3 (day 30), Follow-Up (day 60)
  Change (increase or decrease) in LS-3 total score between baseline and follow-up. Minimum score = 3, maximum score = 9. A higher score indicates more frequent feelings of loneliness.
San Diego Wisdom Scale (SD-WISE) | Baseline (day 1), Follow-Up (day 60)
  Change (increase or decrease) in SD-WISE total score and sub-scores (Acceptance of Divergent Perspectives, Decisiveness, Emotional Regulation, Pro-Social Behaviors, Self-Reflection, Social Advising, and Spirituality) between baseline and follow-up. For the total score and all sub-scores, the minimum score = 1, maximum score = 5. A higher score indicates a better outcome.
Level of Personality Functioning Scale (LPFS) | Baseline (day 1), Time 2 (day 15), Time 3 (day 30), Follow-Up (day 60)
  Change (increase or decrease) in LPFS total score between baseline and follow-up. Minimum score = 12, maximum score = 48. A higher score indicates more severe impairment in personality functioning.
Continuous Performance Test (Full-Length Version) | Baseline (day 1), Time 3 (day 30), Follow-Up (day 60)
  Change (increase or decrease) in CPT scores (Detectability, Omissions, Commissions, Perseverations) between baseline and follow-up.
  CPT scores are calculated as T-Scores (minimum=0, maximum=100). Higher Commission and Perseveration scores indicate a higher level of impulsivity. Higher Detectability, Omission, and Commission scores indicate a higher level of inattentiveness.
Read the Mind in the Eyes Task (RMET). Minimum score = 0, maximum score = 37. Higher score indicates greater accuracy in identifying facial emotion expressions. | Baseline (day 1), Follow-Up (day 60)
  Change (increase or decrease) in RMET score and sub-scores at time 2, time 3, and follow-up, as compared to baseline.
Belmont Emotion Sensitivity Test (BEST) | Baseline (day 1), Follow-Up (day 60)
  Change (increase or decrease) in BEST score for each condition (Happiness, Fear, Anger) at time 2, time 3, and follow-up, as compared to baseline. For each condition, minimum score = 0, maximum score = 56. A higher score indicates greater accuracy in differentiating facial emotion expressions.
Digit Span Test (DST) | Baseline (day 1), Time 2 (day 15), Time 3 (day 30), Follow-Up (day 60)
  Change (increase or decrease) in DST total score and sub-scores (Digits Forward and Digits Backward) at time 2, time 3, and follow-up, as compared to baseline. The DST total score has a minimum of 0 and a maximum of 30. The Digits Forward sub-score has a minimum of 0 and a maximum of 16. The Digits Backward sub-score has a minimum of 0 and a maximum of 14.
  A higher total score indicates greater memory and attention ability. A higher Digits Forward score primarily indicates greater attention/concentration. A higher Digits Backward score primarily indicates better working memory.
Daily Ecological Momentary Assessment (EMA) Measures | Daily, days 1-30
  Trends over time of scores/ratings on all EMA questions and the 1-minute version of the CPT.
  The EMA Measures include:
  * General Functioning: "Did you attend work/school today?" (yes/no) A higher number of days attending work/school indicates better functioning.
  * Social Functioning (# of social interactions since last assessment): Minimum value = 0, no maximum value. A higher number indicates a more active social life.
  * Psychological & Interpersonal States: 14 individual questions, each rated from 0-2. Questions are considered individually, rather than combined into summary scores. A higher score indicates that the participant identifies more strongly with the psychological/interpersonal state (e.g., "I feel securely connected to at least one person I care about." or "I am on alert for signs of rejection.")
  * CPT (1-minute version): The minimum and maximum scores and interpretation of the 1-minute CPT are the same as the full-length version listed above.
Digit Symbol Matching Test (DSMT) | Baseline (day 1), daily days 1-30, Time 3 (day 30), Follow-Up (day 60)
  Changes (increase or decrease) and trends in DSMT score at time 3 and follow up as compared to baseline, and across the 30 days of EMA. The score indicates processing speed.
Client Satisfaction Questionnaire (CSQ-8) | Time 2 (day 15)
  Acceptability measure.

CONTACTS AND LOCATIONS:
Overall Officials: Lois W Choi-Kain, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi-Kain LW, Murray GE, Jurist J, Ren B, Germine L. Online psychoeducation and digital assessments as a first step of treatment for borderline personality disorder: A protocol for a pilot randomized controlled trial. PLoS One. 2023 Dec 7;18(12):e0294331. doi: 10.1371/journal.pone.0294331. eCollection 2023. PMID 38060545